CLINICAL TRIAL: NCT03529305
Title: Effects of Different Frequency rTMS on Brain Functional and Structural Alterations in Stroke Patient: Multi-modal MRI Study
Brief Title: Effects of rTMS on Brain Alterations in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Yating Lv, PhD, Associate Investigator, Hangzhou Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017YFC1310002
Record Dates: First submitted 2018-04-19; First posted 2018-05-18 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Stroke
Keywords: Stroke; rTMS; MRI
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low frequency rTMS (Experimental): Patients receive low frequency rTMS treatment and physical therapy. rTMS is applied over primary motor (M1) cortex of the unaffected side for two weeks, 5 consecutive days each week.
  Interventions: Device: rTMS; Other: Physical therapy
- High frequency rTMS (Experimental): Patients receive high frequency rTMS treatment and physical therapy. rTMS is applied over primary motor (M1) cortex of the affected side for two weeks, 5 consecutive days each week.
  Interventions: Device: rTMS; Other: Physical therapy
- Physical therapy (Active Comparator): Patients receive physical therapy for two weeks.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Device: rTMS — Receive rTMS treatment to the primary motor cortex (M1)
  Arms: High frequency rTMS; Low frequency rTMS
Other: Physical therapy — Receive physical therapy

SUMMARY:
In this study, the investigators aim to evaluate functional and structural improvements in the brain of stroke patients after rTMS treatment using multi-modal MRI techniques. Specifically, the investigators sought to determine whether rTMS treatment modulate the brain function and structure in patients and, if so, whether different frequency of the rTMS treatment will affect the degree of the motor recovery in patients' brain.

The patients will be randomized into three groups: Experimental group 1 (TMS group) received low frequency rTMS; Experimental group 2 (TMS group) received high frequency rTMS; The third group who received only physical therapy constituted the control group. All patients undergo MRI scan one day before and after rTMS treatment.

DETAILED DESCRIPTION:
As the second leading cause of death and major cause of disability in the world, stroke is the rapid loss of brain function due to disturbance in the blood supply to the brain. Approximately two thirds of patients with stroke have impaired motor function even at three to six months after stroke onset. The abnormally increased interhemispheric inhibition driven from the unaffected to the affected hemisphere is associated with the motor impairment, which is characterized by increased cortical excitability in the unaffected hemisphere and decreased cortical excitability in the affected hemisphere. Rebalancing the cortical excitability between two hemispheres is associated with a better overall prognosis.

Repetitive transcranial magnetic stimulation (rTMS) is a painless, noninvasive brain stimulation technique. High-frequency rTMS facilitates cortical excitability, whereas low-frequency rTMS decreases the cortical excitability of the stimulated hemisphere. Therefore, rTMS can be used to increase and decrease the cortical excitability of the affected and unaffected hemispheres, respectively, and may facilitate motor function after stroke. However, the previous studies commonly applied behavioral scales to evaluate the effect of the rTMS treatment, little is known how the brain function and structure recover after rTMS treatment and whether the different frequency of rTMS will affect the recovery in the brain of stroke patients.

Non-invasive neuroimaging techniques provide promising avenues to detect brain function and structure in patients after stroke onset and have been increasingly applied to this disease. The morphology of the brain (cortical thickness, gray matter volume) is commonly assessed using T1-weighted MRI (Structural MRI). Diffusion tensor imaging (DTI) is a promising technique to study human brain structure, especially white matter anatomy, by providing multiple quantitative parameters to characterize tissue microstructure from different aspects. Functional magnetic resonance imaging (fMRI) is a functional neuroimaging technique which measures the changes of the blood oxygenation level-dependent (BOLD) signal that are highly correlated with neural activities. Task fMRI which applies stimulus-response pattern to identify the regions activated by performance of a cognitive task, while resting-state fMRI (rs-fMRI) is a promising tool to map intrinsic function of the human brain, which has unique advantages in clinical conditions because it does not require participants to engage in cognitive activities.

In this study, the investigators aim to evaluate functional and structural improvements in the brain of stroke patients after rTMS treatment using multi-modal MRI techniques. Specifically, the investigators sought to determine whether rTMS treatment modulate the brain function and structure in stroke patients and, if so, whether different frequency of the rTMS treatment will affect the degree of the motor recovery in patients' brain.

ELIGIBILITY:
Inclusion Criteria:

1. First-ever ischemic stroke
2. One to six months after stroke onset;
3. Mini Mental State Examination (MMSE) score > 24;
4. Brunnstrom recovery stage (BRS) for hand fingers of 3-5
5. Motor deficits of the unilateral upper limb

Exclusion Criteria:

Patients with hemorrhage, leukoaraiosis, epilepsy, migraine or psychiatric diseases history are excluded in this study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain functional changes after rTMS treatment | One day before and after two weeks' treatment
  Brain functional changes in patients' brain measured by fMRI
Brain morphological changes after rTMS treatment | One day before and after two weeks' treatment
  Gray matter morphological changes in patients' brain measured by high resolution T1-weighted MRI
Brain structural changes after rTMS treatment | One day before and after two weeks' treatment
  White matter anatomical changes in patients' brain measured by DTI

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Feng Zang, MD, Principal Investigator — Hangzhou Normal University
Locations (2):
- China (2):
  - Affiliated Hospital of Nanjing University of Chinese Medicine, Nanjing, Jiangsu
  - Hangzhou Normal University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided